CLINICAL TRIAL: NCT06104007
Title: Safety and Efficacy of Paclitaxel Coated PTCA Balloon Catheter With a Shellac Plus Vitamin E Excipient (GENOSS® DCB) in Patients With Coronary In-stent Restenosis (ISR): A Prospective, Multi-center, Observational Study
Acronym: SFRGENISTA
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Bon-Kwon Koo, Professor, Seoul National University Hospital
Other Study IDs: 2304-037-1420
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Coronary Artery Disease; In-stent Restenosis
Keywords: Coronary Artery Disease; In-stent Restenosis; Drug-coated Balloon
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Genoss® DCB: Patients with coronary in-stent restenosis (ISR) who underwent percutaneous coronary intervention using the Genoss® DCB
  Interventions: Device: Genoss® DCB

INTERVENTIONS:
Device: Genoss® DCB — This study includes patients with coronary in-stent restenosis (ISR) who have undergone percutaneous coronary intervention (PCI) according to standard treatment protocols using the Genoss® DCB and have agreed to participate in the clinical research. The decision on which drug-coated balloon (DCB) to use during PCI is entirely based on the patient's condition and the characteristics of the coronary lesions identified through angiography. Thus, it's not possible to determine in advance to use the Genoss® DCB before the procedure, nor can the number of drug-coated balloon catheters to be used during the procedure be known or decided upon beforehand.

SUMMARY:
The SFRGENISTA study aims to evaluate the long-term efficacy and safety of a paclitaxel-coated balloon catheter containing shellac and vitamin E excipients (Genoss® DCB) in patients with coronary in-stent restenosis (ISR).

DETAILED DESCRIPTION:
Drug-coated balloon (DCB) treatment is a therapeutic strategy to overcome in-stent restenosis (ISR) that occurs after drug-eluting stent (DES) implantation. The 2018 European guidelines on myocardial revascularization recommend DCB treatment in patients with bare-metal stent (BMS) or DES ISR lesions. The Sequent Please World Wide Registry has shown that DCB therapy is safe and exhibits a low target lesion revascularization (TLR) rate in a large population.

The Genoss® DCB is coated with 3µg/mm² of paclitaxel along with shellac, a hydrophilic excipient for rapid release and diffusion into the tissue. Additionally, it incorporates vitamin E, an antioxidant known to directly prevent the accumulation of smooth muscle cells associated with neointimal hyperplasia that arises from the vessel wall being damaged by the balloon catheter. The catheter was designed to enhance trackability and pushability, minimize vascular damage with the application of a hydrophilic coating to the distal part, and use a soft yet durable end-tip for easier access to the target lesion. In a clinical trial comparing Genoss® DCB to the Sequent® Please (B-BRAUN) DCB, the in-segment late lumen loss at six months after DCB was comparable, and the rates of adverse clinical events were similar.

Given this background, this study intends to investigate the long-term efficacy and safety of the Genoss® DCB in patients with coronary ISR.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary in-stent restenosis (ISR) who underwent percutaneous coronary intervention using the Genoss® DCB.
* Participants who have agreed to the clinical trial protocol and the clinical follow-up study plan, voluntarily decided to participate in this clinical research, and have provided written consent on the research participant agreement form.

Exclusion Criteria:

* Women of childbearing age who plan to become pregnant during the study duration.
* Patients scheduled for a surgery within 12 months of enrollment that requires discontinuation of antiplatelet agents.
* Patients for whom the expected remaining life span is less than one year.
* Patients who presented with cardiogenic shock at the time of their visit and, based on medical assessment, are predicted to have a low likelihood of survival.
* Patients currently involved in a randomized medical device study.
* Patients deemed by the researcher to be unsuitable for this study or whose participation might increase associated risks.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary in-stent restenosis who underwent percutaneous coronary intervention using the Genoss® DCB.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Target lesion failure | 1 year
  A composite of cardiac death, target vessel myocardial infarction, and target lesion revascularization

SECONDARY OUTCOMES:
Major adverse cardiac event | 1 year
  A composite of cardiac death, myocardial infarction, and revascularization
All-cause death | 1 year
  All-cause death
Cardiac death | 1 year
  Cardiac death
Myocardial infarction | 1 year
  Myocardial infarction
Target vessel myocardial infarction | 1 year
  Target vessel myocardial infarction
Revascularization | 1 year
  Revascularization
Ischemic driven target lesion revascularization | 1 year
  Ischemic driven target lesion revascularization
Major bleeding (BARC type 3, 5) | 1 year
  Major bleeding (BARC type 3, 5)
Stroke | 1 ye
  Stroke
Acute stent thrombosis (within 24 hours), subacute stent thrombosis (within 30 days), late stent thrombosis (within 1 year) | 1 year
  Acute stent thrombosis (within 24 hours), subacute stent thrombosis (within 30 days), late stent thrombosis (within 1 year)

CONTACTS AND LOCATIONS:
Locations (1):
- Bon-Kwon Koo, Seoul, South Korea